CLINICAL TRIAL: NCT00598611
Title: An Exploratory Phase III, Randomised, Double-blind, Therapeutic Single Dose-related Effect, Parallel Group Study to Assess and Compare the Effects of 5 mg vs. 20 mg Desloratadine on Skin Lesions in Patients With Chronic Urticaria (CU)
Brief Title: Effects of 5 mg vs. 20 mg Desloratadine on Skin Lesions in Patients With Chronic Urticaria (CU)
Acronym: AUD2OCU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Essex Pharma GmbH (Industry)
Responsible Party: Principal Investigator, K. Weller, Dr. Karsten Weller, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P04805-V2.0; EudraCT number: 2006-003686-13
Record Dates: First submitted 2008-01-10; First posted 2008-01-22 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Urticaria
Keywords: urticaria
MeSH Terms: conditions — Chronic Urticaria; Urticaria | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): desloratadine 20 mg
  Interventions: Drug: desloratadine
- 2 (Active Comparator): desloratadine 20 mg
  Interventions: Drug: desloratadine

INTERVENTIONS:
Drug: desloratadine — singel dose, oral, 20 mg
  Arms: 1
Drug: desloratadine — single dose, oral, 5 mg
  Arms: 2

SUMMARY:
The purpose of this study is to compare urticaria lesions (size, kinetics) by thermography, volumetry and digital time lapse photography in CU patients treated with desloratadine 5 mg or desloratadine 20 mg. Hypothesis: Updosing of desloratadine (20mg) is more efficient in the treatment of urticarial lesions as compared to standard dosing (5 mg desloratadine).

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with moderate to severe CU for more than 6 weeks. Urticaria symptoms must comprise wheal and itch.
2. Patients must exhibit spontaneous urticaria lesions in the randomization visit.
3. History of beneficial effects of antihistaminic treatment.
4. Age between 18 and 60 years.
5. Female patients must be using adequate contraceptive precautions (highly effective method), or they must be postmenopausal, surgically sterilised, or hysterectomised (for details please see protocol).
6. Female patients must be using adequate contraceptive precautions (contraceptive pill, depot, double barrier methods), or they must be postmenopausal, surgically sterilised, or hysterectomised.
7. Voluntarily signed written informed consent.

Exclusion Criteria:

1. The presence of permanent severe diseases, especially those affecting the immune system, except CU.
2. The presence of permanent gastrointestinal condition which may influence the oral therapy (chronic diarrhea diseases, congenital malformations or surgical mutilations of the gastrointestinal tract).
3. History or presence of epilepsy, significant neurological disorders, cerebrovascular attacks or ischemia.
4. History or presence of myocardial infarction or cardiac arrhythmia which requires drug therapy.
5. Evidence of severe renal dysfunction
6. Evidence of significant hepatic disease (liver enzymes twice the upper reference value).
7. The presence of galactose intolerance, lapp lactase deficiency or glucose galactose malabsorption.
8. History of adverse reactions including hypersensitivity to DL and Loratadine.
9. Intake of medicaments that could cause QT changes (drugs listed on www.qtdrugs.org).
10. Presence of active cancer which requires chemotherapy or radiation therapy.
11. Presence of acute urticaria / angioedema including laryngeal edema
12. History or presence of alcohol abuse or drug addiction.
13. Participation in any clinical trial within 4 weeks prior to enrolment.
14. Intake of oral corticosteroids or other immunosuppressive therapy within 14 days prior to the beginning of the study.
15. Use of depot corticosteroids or chronic systemic corticosteroids within 21 days before beginning of the study.
16. Pregnancy or breast-feeding.
17. Existing or planned placement in an institution after ruling according to § 40 passage 1 number 4 AMG (Arzneimittelgesetz).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Reduction in size of existing spontaneous urticaria lesions (wheal and flare) as assessed by thermography. | 5 hours

SECONDARY OUTCOMES:
Reduction in size of existing spontaneous urticaria lesions (wheal and flare) as assessed by volumetry and digital time lapse photography. | 5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, MD, Principal Investigator — Allergie-Centrum-Charite
Locations (1):
- Allergie-Centrum-Charite, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Weller K, Ardelean E, Scholz E, Martus P, Zuberbier T, Maurer M. Can on-demand non-sedating antihistamines improve urticaria symptoms? A double-blind, randomized, single-dose study. Acta Derm Venereol. 2013 Mar 27;93(2):168-74. doi: 10.2340/00015555-1434. PMID 23053062
- See also: Related Info — http://www.urtikaria.net